CLINICAL TRIAL: NCT05657418
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics of JS107 in Patients With Advanced Pancreatic Cancer
Brief Title: A Clinical Study to Evaluate the Safety and Tolerability of JS107 in Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company research and development strategy adjustment
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS107-002-I
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: Sequential
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS107 (Experimental)
  Interventions: Drug: JS107
- JS107 combination with Toripalimab (Experimental)
  Interventions: Combination Product: JS107 combination with Toripalimab

INTERVENTIONS:
Drug: JS107 — JS107, i.v., q3w
  Arms: JS107
Combination Product: JS107 combination with Toripalimab — JS107 i.v., q3w combine with Toripalimab
  Arms: JS107 combination with Toripalimab

SUMMARY:
The purpose of this phase I clinical study was to evaluate the safety and tolerability of JS107 monotherapy and combination with Toripalimab in patients with Advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study with full informed consent and signed written informed consent form;
2. Aged ≥18 years and ≤75 years when the subject signed the informed consent;
3. Locally advanced unresectable or metastatic malignant solid tumors diagnosed histologically ;
4. Provide past tumor samples or fresh tumor tissue biopsy samples;
5. The physical status score is 0 or 1 on the Eastern Oncology Collaboration (ECOG) scale;
6. The expected survival is ≥3 months;
7. There should be at least one measurable lesion according to RECIST V1.1 evaluation criteria;
8. Any adverse events and/or complications resulting from prior treatment, including surgery or radiation therapy, that have been adequately resolved to level 0 or 1 (according to the NATIONAL Cancer Institute Standard for General Terminology of Adverse Events (NCI-CTCAE 5.0) or to the level specified in the inclusion criteria; Any grade of hair loss/pigmentation and other long-term toxicity caused by treatment, except those that are irreversible and do not affect study dosing/compliance and patient safety at the discretion of the investigator;
9. Good organ function；
10. Within 7 days prior to the first dose, women of reproductive age must be confirmed as having a negative serum pregnancy test and consent to use effective contraception during the duration of study drug use and for 6 months after the last dose. Male patients with a female partner of reproductive age agreed to use effective contraception during the study drug use period and for 6 months after the last dose.

Exclusion Criteria:

1. Prior treatment with drugs or other therapies targeting CLDN18.2;
2. A history of severe allergic reactions to to any component of JS107;
3. Received radiotherapy (except palliative radiotherapy for symptom control), chemotherapy, targeted therapy, endocrine therapy and other antitumor therapies, or other investigational drugs within 4 weeks before the administration of the first dose;
4. Received any monoclonal antibody or antibody conjugate within 4 weeks prior to administration of the first study drug or within 5 half-lives (depend on whichever is shorter);
5. Serious infection (CTCAE> grade 2) occurred within 14 days before the first dose;
6. Patients with other malignant tumors except for the tumor treated in the study within 5 years prior to the administration of the first study drug (exceptions included: cured malignancies that had not recurred within 3 years prior to study enrollment; Completely resected basal and squamous cell skin cancers; Complete resection of any type of carcinoma in situ, etc.);
7. Major organ surgery was performed or significant trauma was present within 4 weeks before the first administration of the study drug;
8. Weight loss 10% within 2 months before drug administration, or other indicators of severe malnutrition, or body mass index (BMI)<17.5 at the time of signing the informed consent.
9. The following conditions were present within 6 months prior to the first study dose: myocardial infarction, severe/unstable angina, NYHA class 2 or higher cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestive heart failure , hypertensive crisis, or hypertensive encephalopathy; patients with known hypertension, coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must be treated with optimal stabilization as determined by the treating physician medical plan;
10. Pericardial effusion, pleural effusion or abdominal effusion with clinical symptoms, signs or requiring symptomatic treatment;
11. Poorly controlled pain related;
12. The presence of uncontrolled or symptomatic active central nervous system (CNS) metastases, which can be manifested by the onset of clinical symptoms, cerebral edema, spinal cord compression, carcinomatous meningitis, leptomeningeal disease, and/or progressive growth;
13. Active infection, including tuberculosis (clinical diagnosis including clinical history, physical examination and imaging findings, as well as TB tests according to local medical routine), hepatitis B, hepatitis C or human immunodeficiency virus (HIV antibody positive);
14. Pregnant or lactating women;
15. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
16. Have serious psychological or mental abnormality, which affects the compliance of the subject to participate in this clinical study;
17. Idiopathic pulmonary fibrosis, drug-induced pneumonia, machine-induced pneumonia (bronchiolitis obliterans), radioactive pneumonia with clinical symptoms or requiring steroid treatment, active pneumonia, or other moderate to severe lung diseases that seriously affect lung function ;
18. History of autoimmune disease;
19. Persons who have an immunodeficient disease or the other chronic immunosuppressive therapy, or who have received systemic immunomodulatory drugs (including, but not limited to, interferon or IL-2) within 14 days before first dose or within the 5 half-life of the drug (depend on whichever is longer), or received systemic glucocorticoid therapy (10mg daily of prednisone or equivalent glucocorticoids) or other systemic immunosuppressive therapy within 14 days before first dose;
20. Received any live vaccine (e.g. influenza vaccine against infectious diseases, chickenpox vaccine, etc.) within 14 days before first dose;
21. Other conditions deemed inappropriate for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
MTD | Up to approximately 12 months from first patient in.
  Determine maximum tolerated dose (MTD, if possible)
RP2D | Up to approximately 24 months from first patient in.
  Recommended phase II dose (RP2D) for JS107 monotherapy and combination therapy

SECONDARY OUTCOMES:
Drug concentrations in plasma | Up to approximately 24 months from first patient in.
  Drug concentrations in individual subjects at different time points after dosing
Immunogenicity | Up to approximately 24 months from first patient in.
  Incidence of anti-drug antibody (ADA) and/or neutralizing antibody (Nab), titer of ADA positive samples
ORR | Up to approximately 24 months from first patient in.
  Objective response rate (ORR) was assessed based on RECIST V1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No